CLINICAL TRIAL: NCT02160210
Title: Ultrafine Endoscope for Unsedated Colonoscopy is an Effective Method to Reduce Abdominal Pain:a Prospective Randomized Study.
Brief Title: Ultrafine Endoscope for Colonoscopy in Diagnosis of Colorectal Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Youlin Yang ,MD (Other)
Responsible Party: Sponsor-Investigator, Youlin Yang ,MD, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-001
Record Dates: First submitted 2014-06-09; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Colon Disease;; Rectal Disease
MeSH Terms: conditions — Colonic Diseases; Rectal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrafine Endoscope (Experimental): The ultrafine endoscope for colonoscopy with water method is performed in screening the colorectal diseases.
  Interventions: Device: Ultrafine Endoscope

INTERVENTIONS:
Device: Ultrafine Endoscope — Ultrafine endoscope reaching to the cecum within 15mins is thought to be successful.Water colonoscopy with standard colonoscope will be performed in unsuccessful subjects subsequently.
  Other Names: Transnasal gastroscope

SUMMARY:
This study is the evaluation of ultrafine endoscope (with small caliber and turning radius )for colonoscopy in decreasing abdominal pain of patients . 60 patients will be accepted in this trial.

DETAILED DESCRIPTION:
The aim of this study is to investigate the advantages of an endoscope with smaller turning radius and softer insert section in reducing patients' abdominal pain in colonoscopy. Transnasal gastroscope was selected in this study , because of its small caliber (5.9mm) and small turning radius . Visual analogue scale(VAS),cecum intubation time and cecum intubation rate were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnostic colonoscopy;
2. Subjects able to provide informed consent

Exclusion Criteria:

1. Patients with poor bowel preparation;
2. Contraindications of the colonoscopy;
3. Prior partial or complete colectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
VAS abdominal pain scores | up to two months
  VAS abdominal pain scores include pain scores in the insertion phase of splenic flexure,hepatic flexure,and ileocecal junction.(0=no pain and 10=most severe pain imaginable).

SECONDARY OUTCOMES:
Cecum intubation time | up to two months
  Insertion time from rectum to reach the cecum.
The time to reach the splenic flexure | up to two months
  Insertion time from rectum to reach the flexure.
The time to reach the hepatic flexure | up to two months
  Insertion time from rectum to hepatic flexure.
The success rate of the cecal intubation within 15 minutes | up to two months
  Percentage of successful colonoscopy (insertion of ultrafine endoscope into cecum within 15 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Youlin Yang, MD, Principal Investigator — Gastroenterology Department of The 1st Affiliated Hospital of Harbin Medical University
Locations (1):
- The Gastroenterology Department of The 1st Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China